CLINICAL TRIAL: NCT06019455
Title: A Prospective Observational Study on the Level of Patient Participation in Lung and Esophageal Cancer Patients Treated With Definitive Radiochemotherapy.
Brief Title: The Level of Patient Participation in Lung and Esophageal Cancer Patients Treated With Definitive Radiochemotherapy.
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Other Study IDs: 2023-FXY-017
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Esophageal Cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: Patients undergoing definitive radiochemotherapy ± immunotherapy will be assessed about the level of participation in their medical processes.

SUMMARY:
This study aims to assess the level of participation of thoracic cancer patients undergoing definitive radiotherapy and chemotherapy ± immunotherapy in their medical processes and the association between the level of participation and patients' side effects, quality of life, and long-term survival. Additionally, this study will rate the level of participation from both the patients' and medical staff's perspectives and will compare the differences in ratings from these two viewpoints, as well as their impact on treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced non-small cell lung cancer, limited-stage small cell lung cancer, and esophageal cancer.
* Planned to undergo definitive chemoradiotherapy ± immunotherapy;
* Males or females aged 18 to 75;
* Able to communicate with medical staff.

Exclusion Criteria: Patients with cognitive impairments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced non-small cell lung cancer, limited-stage small cell lung cancer, or esophageal cancer
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of >=Grade 3 toxicities | 2 years
  The percentage of patients who develop >=Grade 3 toxicities

SECONDARY OUTCOMES:
Overall survival | 2 years
  2-year survival rate
Progression-free survival | 2 years
  2-year progression-free survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided